CLINICAL TRIAL: NCT02160548
Title: Effect of Adding Nebulized Salbutamol to Intravenous Atropine and Oxygen During Resuscitation of OP Pesticide Poisoned Patients
Brief Title: Adding Nebulized Salbutamol to Intravenous Atropine and Oxygen in OP Poisoning
Acronym: SalbutamolOP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sylhet M.A.G.Osmani Medical College (Other)
Collaborators: University of Edinburgh (Other)
Responsible Party: Principal Investigator, Dr. Fazle Rabbi Chowdhury, Consultant, Medicine, Sylhet M.A.G.Osmani Medical College
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Medicine SOMCH
Record Dates: First submitted 2014-06-07; First posted 2014-06-10 (Estimated); Last update posted 2015-12-29 (Estimated); Status verified 2015-12

CONDITIONS: Organophosphate Poisoning
Keywords: Organophosphate, insectiside, Salbutamol, Atropine
MeSH Terms: conditions — Organophosphate Poisoning | interventions — Standard of Care; Atropine; pralidoxime; Albuterol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 'Standard care' (Placebo Comparator): Standard care= Intravenous fluids, Oxygen by face mask, Intubation if necessary, Mechanical ventilation (Engstrom Pro by GE) if necessary, Cardiac monitor (Infunix IP4050), Atropine (anti-muscarinic drug; G-Atropine) by intravenous route, Pralidoxime (acetylcholinesterase reactivating oxime drug; PAM-A) by intravenous route.
  Interventions: Drug: Standard care
- 'Standard care+ 2.5 mg Salbutamol' (Experimental): Standard care+ 2.5 mg Salbutamol= Nebulized salbutamol (Ventolin respiratory solution) 2.5 mg stat and once only with standard care
  Interventions: Drug: Standard care+ 2.5 mg Salbutamol
- 'Standard care+ 5 mg Salbutamol' (Experimental): Standard care+ 5 mg Salbutamol= Nebulized salbutamol (Ventolin respiratory solution) 5 mg stat and once only with standard care
  Interventions: Drug: Standard care+ 5 mg Salbutamol

INTERVENTIONS:
Drug: Standard care — Standard management for OP poisoning
  Other Names: Intravenous fluids; Intubation if necessary,; Mechanical ventilation if necessary (Engstrom Pro); Atropine (anti-muscarinic; G-Atropine); Pralidoxime (acetylcholinesterase reactivating oxime; PAM-A); Oxygen by face mask by intravenous route,
  Arms: 'Standard care'
Drug: Standard care+ 2.5 mg Salbutamol — Ventolin respiratory solution 2.5 mg
  Other Names: Ventolin
  Arms: 'Standard care+ 2.5 mg Salbutamol'
Drug: Standard care+ 5 mg Salbutamol — Ventolin respiratory solution 5 mg
  Other Names: Ventolin
  Arms: 'Standard care+ 5 mg Salbutamol'

SUMMARY:
We hypothesize that salbutamol will speed removal of alveolar fluid compared to atropine alone in OP poisoned patients. We propose to compare the effect of two stat doses of nebulized salbutamol (2.5 mg; 5.0 mg), with nebulized saline placebo, in symptomatic patients receiving standard resuscitation with atropine, oxygen, and fluids after poisoning with OP pesticides. 25 patients will be randomised to each arm (total 75 patients). Primary outcome will be oxygen saturation's over the following 60 min during resuscitation. Secondary outcomes will include atropine dose administered, speed to stabilization, aspiration or pneumonia, intubation, tachydysrhythmias, and mortality. A positive outcome will result in design of a large definitive phase III study.

DETAILED DESCRIPTION:
Pesticide self-poisoning kills over 300,000 people every year (1). Most deaths occur in rural Asia where widespread use of pesticides to boost food production allows easy access at stressful times. The WHO now recognizes pesticide poisoning to be the single most important global means of suicide (2) Amongst pesticides, organophosphorus (OP) and carbamate insecticides are of most concern, causing about 2/3 of deaths (1,3). These insecticides inhibit the enzyme acetylcholinesterase (AChE), producing an 'acute cholinergic crisis' with reduced consciousness, bradycardia, hypotension, and acute respiratory failure. On arrival at hospital, patients are resuscitated with atropine and, for OPs, an oxime AChE reactivator (4). Unfortunately, this treatment is often inadequate and many still die (5). A recent Bangladeshi RCT showed that rapid resuscitation of patients with atropine saves lives (6). This study compared a faster 'doubling dose' method of atropinisation with a standard bolus method during resuscitation. It reported quicker stabilisation and a 14% absolute reduction in mortality.

Rationale: Atropine only stops production of fluid and does not speed its removal from the lung. Therefore a treatment that increases removal, to complement atropine-induced cessation of production, could reduce fluid in the lungs and speed return effective oxygen exchange. A single nebulised dose of the beta-adrenergic agonist salbutamol may increase removal since it increases alveolar fluid removal via the epithelial sodium channel. A pilot clinical study is required to test the hypothesis and to provide data for powering a large phase III RCT.

Research question: Will addition of the beta-adrenergic agonist salbutamol to atropine during resuscitation improve oxygenation, reduce the need for atropine, and speed stabilisation?

Objectives:General Objectives: To test the efficacy of salbutamol at increasing oxygenation and speeding resuscitation.

Specific Objectives: To test whether salbutamol alters dose of atropine administered and incidence of tachydysrhythmias.

Total duration of the study will be one year and all patients aged 12 years or older with clinical features of OP/carbamate poisoning requiring oxygen and atropine will be enrolled. The study will be done in three arms.

ELIGIBILITY:
Inclusion Criteria:

* age 12 yrs or older
* clinical features of OP poisoning
* requiring oxygen and atropine and give consent

Exclusion Criteria:

* age 11 yrs or younger
* no requirement for atropine

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2015-04; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Improvement of oxygen saturation | 60 minutes
  Improvement of oxygen saturation from the base line to normal level after adding nebulized salbutamol to regular I/V atropine and oxygen therapy.

SECONDARY OUTCOMES:
Heart rate, respiratory rate and Blood pressure | 60 minutes
  Settlement of heart rate, respiratory rate and blood pressure to normal range after adding salbutamol to regular management.

OTHER OUTCOMES:
Atropine dose | 120 minutes
  Requirement of total atropine dose until full atropinization (before put in to maintenance dose) after adding nebulized salbutamol

CONTACTS AND LOCATIONS:
Overall Officials: Fazle R Chowdhury, FCPS, Principal Investigator — Consultant, Medicine, Sylhet M.A.G.Osmani Medical Collge, Sylhet, Bangladesh; Michael Eddleston, PhD, Principal Investigator — Professor of Clinical Toxicology, University of Edinburgh
Locations (1):
- Sylhet M.A.G.Osmani Medical College Hospital, Sylhet, Sylhet Division, Bangladesh

REFERENCES:
- [Background] Abedin MJ, Sayeed AA, Basher A, Maude RJ, Hoque G, Faiz MA. Open-label randomized clinical trial of atropine bolus injection versus incremental boluses plus infusion for organophosphate poisoning in Bangladesh. J Med Toxicol. 2012 Jun;8(2):108-17. doi: 10.1007/s13181-012-0214-6. PMID 22351300
- [Background] Eddleston M, Buckley NA, Eyer P, Dawson AH. Management of acute organophosphorus pesticide poisoning. Lancet. 2008 Feb 16;371(9612):597-607. doi: 10.1016/S0140-6736(07)61202-1. PMID 17706760
- [Background] Gunnell D, Eddleston M, Phillips MR, Konradsen F. The global distribution of fatal pesticide self-poisoning: systematic review. BMC Public Health. 2007 Dec 21;7:357. doi: 10.1186/1471-2458-7-357. PMID 18154668
- [Background] Eddleston M. Patterns and problems of deliberate self-poisoning in the developing world. QJM. 2000 Nov;93(11):715-31. doi: 10.1093/qjmed/93.11.715. PMID 11077028